CLINICAL TRIAL: NCT00193583
Title: A Phase I Study of Weekly Topotecan in Combination With Carboplatin in Two Different Schedules for Patients With Refractory and/or Advanced Solid Tumors
Brief Title: Weekly Topotecan in Combination With Carboplatin in Two Different Schedules for Refractory and/or Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: SCRI Oncology Research Consortium, SCRI
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI REFMAL 40; 104864-707
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2011-05-04 (Estimated); Status verified 2011-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Topotecan; Carboplatin

INTERVENTIONS:
Drug: Topotecan
Drug: Carboplatin

SUMMARY:
In this phase I study we will characterize the safety, tolerability, maximum tolerated dose and dose-limiting toxicity of weekly bolus topotecan when administered in combination with two different dosing schedules of carboplatin. We will also evaluate any antitumor activity of these combination regimens.

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be receive:

* Topotecan + Carboplatin

In order to determine the most appropriate dosing regimen to progress into future phase II trials, two different dosing schedules of topotecan and carboplatin will be utilized (ARM I and ARM II). Patients will be accrued to both treatment arms simultaneously.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Adult patients at least 18 years old
* Advanced solid tumors refractory to conventional therapy
* ECOG performance status must be 0 or 1
* Patients may have received no more than 3 prior chemotherapy regimens
* Adequate bone marrow, liver and kidney function
* Able to understand the nature of the study and give written informed consent.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Active concurrent infections or serious underlying medical conditions
* Known HIV positivity
* Female patients who are pregnant or lactating
* Received both topotecan and carboplatin

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2003-05; Primary Completion 2004-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose

SECONDARY OUTCOMES:
Dose limiting toxicity
All over response

CONTACTS AND LOCATIONS:
Overall Officials: Howard A. Burris, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (1):
- Tennessee Oncology, PLLC, Nashville, Tennessee, United States